CLINICAL TRIAL: NCT06119308
Title: Pilot of a Brief Cognitive Behavioral Therapy Intervention to Enhance Benzodiazepine Deprescribing in Older Adults
Brief Title: Brief Cognitive Behavioral Therapy to Enhance Benzodiazepine Deprescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of California, San Francisco (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000382
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Benzodiazepine Use; Insomnia; Anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benzodiazepine Medication Taper with Cognitive Behavioral Therapy (Experimental): Brief Cognitive Behavioral Therapy to Enhance Benzodiazepine Deprescribing
  Interventions: Other: Benzodiazepine Medication Taper with Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Benzodiazepine Medication Taper with Cognitive Behavioral Therapy — Brief Cognitive Behavioral Therapy to Enhance Benzodiazepine Deprescribing (led by pharmacist/clinician/psychologist) over a 10-week Trial.

SUMMARY:
The goal of this clinical trial is to conduct a single-arm pilot trial of a brief cognitive-behavioral therapy-enhanced benzodiazepine deprescribing intervention in 20 older adults (aged ≥55 years) prescribed chronic benzodiazepines by their primary care clinicians.

DETAILED DESCRIPTION:
Nearly 10% of Americans aged 55 years and older fill benzodiazepine (BZD) prescriptions annually. Chronic use of BZD place older adults at an increased risk of falls, cognitive impairment, functional decline, preventable hospitalizations, and mortality.

Research study investigators will conduct a single-arm pilot trial of the intervention in 20 adults aged 55 and older currently taking chronic BZDs. The aim is to evaluate feasibility/acceptability of the refined deprescribing intervention using mixed methods. At intervention end, research study investigators will conduct surveys and qualitative interviews with participants to obtain feedback on participant experience and intervention components (e.g., acceptability, usefulness, relevance, satisfaction) as well as views on future format options. Using these data and the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework, research study investigators will further refine the intervention in preparation for larger scale testing and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed chronic benzodiazepines by their primary care clinicians at a Beth Israel Deaconess Medical Center (BIDMC) Primary Care Clinic.

Exclusion Criteria:

* Primary Care Practitioner (PCP) opt out
* Severe anxiety or depression symptoms

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
Feasibility: Retention | Immediately after 10 weeks of participation
  Recruitment, retention (<10% dropout)
Feasibility: Intervention adherence | Immediately after 10 weeks of participation
  Intervention adherence (>75% in at least 2 of 3 sessions)
Acceptability: Open-ended qualitative interview | Immediately after 10 weeks of participation
  Usefulness in supporting tapering process, use of specific skills and mindfulness techniques, clarity/length of sessions, helpfulness, plans to continue, suggestions for improvements, alternative session formats using open-ended qualitative interview.
Change in Benzodiazepine Use | From enrollment to end of intervention at 10 weeks.
  Patient-reported benzodiazepine medication doses with change measured by % change from baseline dose.
Change in Sleep Disturbance Scores | From enrollment to end of intervention at 10 weeks.
  PROMIS Sleep Short Form 8b survey.
Change in Anxiety Scores | From enrollment to end of intervention at 10 weeks.
  PROMIS Anxiety Short Form 8a Survey.

SECONDARY OUTCOMES:
Behavior: Self-efficacy measured by 7-point Likert scale questions | Week 0 and Immediately after 10 weeks of participation
  7-point Likert scale questions: I am confident I can: reduce my benzodiazepine dose; manage anxiety and/or insomnia without medications.
Behavior: Intentions on tapering measured by a 15-point validated scale | Week 0 and Immediately after 10 weeks of participation
  15-point validated measure to assess one's choice predisposition (leaning) towards an option: In the future I will avoid benzodiazepine medications for sleep/anxiety (1=no, 8=unsure, 15=yes)
Behavior: Attitudes on benzodiazepine use measured by 7-point Likert scale | Week 0 and Immediately after 10 weeks of participation
  7-point Likert scale: Reducing benzodiazepine use is: necessary-unnecessary; beneficial-harmful; high-priority-low-priority; worthless-useful.
Behavior: Knowledge on benzodiazepine risk/benefits measured by true/false questions | Week 0 and Immediately after 10 weeks of participation
  Knowledge on benzodiazepine risks/benefits will be assessed with 8 True/False questions
Behavior: Norms of using benzodiazapine medications measured by 7-point Likert Scale | Week 0 and Immediately after 10 weeks of participation
  Using benzodiazepines for sleep/anxiety: risky-safe; beneficial-harmful; pleasant-unpleasant; My doctor/family think(s) I should use benzodiazepines. There are effective treatments for sleep/anxiety other than medications.
Sustainability of Intervention Effect measured by electronic health record review | Up to 6 months post intervention
  Sustainability of benzodiazepine dose reduction, identified by electronic health record review at 3 and 6 months following tapering program completion

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Yeh, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States